CLINICAL TRIAL: NCT02155699
Title: Exercise and Markers of Medial Temporal Health in Youth at Ultra High-risk for Psychosis
Brief Title: Exercise and Markers of Medial Temporal Health in Youth At-risk for Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of Colorado, Denver (Other); National Institute of Mental Health (NIMH) (NIH); Northwestern University (Other)
Responsible Party: Principal Investigator, Vijay Mittal, Assistant Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CU 14-0200; 4R33MH103231-03 (NIH)
Record Dates: First submitted 2014-05-30; First posted 2014-06-04 (Estimated); Results first posted 2024-03-13 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Attenuated Psychosis Syndrome
Keywords: UHR, Remediation, Exercise, Intervention, Psychosis
MeSH Terms: conditions — Motor Activity; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise 1 (Experimental): 65% of V02 Max, 3x per week, 3 months
  Interventions: Behavioral: Exercise 1
- Exercise 2 (Experimental): 85% of VO2 Max, 2x per week, 3 months
  Interventions: Behavioral: Exercise 2
- Waitlist (No Intervention): Waitlist (three months)

INTERVENTIONS:
Behavioral: Exercise 1 — 65% of VO2max and 2 sessions per week
  Arms: Exercise 1
Behavioral: Exercise 2 — 85% intensity and 3 sessions per peek
  Arms: Exercise 2

SUMMARY:
The goal of this proposal is to test the feasibility and effectiveness of cardiovascular exercise in promoting brain health and improving related symptoms (e.g., hearing sounds that are not there, feeling emotionally detached from self and others), cognitive difficulties (troubles with memory and learning), and every day social-occupational functioning in youth at imminent risk for developing a psychotic disorder such as schizophrenia. Understanding how exercise may protect or improve the health of a brain area that is implicated as a major contributing factor to the onset of psychosis may lead to a path-breaking new intervention that does not suffer from many of the side effects, costs, and other barriers that characterize treatments that are currently available for this group. Because a significant portion of high-risk youth go on to develop a psychotic disorder in a short period, intervening at this stage may help to improve the clinical course and ultimately prevent the onset of a devastating and prevalent mental illness.

DETAILED DESCRIPTION:
Accumulating evidence from the animal literature, healthy populations, and schizophrenia studies suggests that regular exercise positively affects integral functions such as neurogenesis, synaptic plasticity and cognition. Likewise, preliminary evidence suggests that aerobic activity has been associated with improved quality of life and a lower level of symptoms in patients with schizophrenia. Because exercise has been found to stimulate human medial temporal neurogenesis, and related abnormalities have been widely observed in studies of schizophrenia, physical activity may be in an important intervention. During the psychosis prodrome, a period immediately proceeding formal onset of psychotic disorders, adolescents experience subtle attenuated symptoms coupled with cognitive deterioration and a global decline in socio-occupational functioning and anywhere between 10-35% go on to transition to a psychotic disorder such as schizophrenia in a two-year period. Despite the promise of exercise interventions, and the critical role medial temporal lobe abnormalities play in etiological models of psychosis, there have been no experimental studies of aerobic exercise in ultra-high risk youth (UHR). Understanding the potential benefits of aerobic exercise in UHR youth is integral as the prodrome is a viable period of intervention in which considerable brain development is still occurring. Further, as there have been challenges associated with many of the available interventions, and an increasing level of potential found in neuroplasticity-based interventions, understanding the effect of exercise on respective brain-behavior holds considerable promise. Experimental research is sorely needed to determine if prescribed aerobic exercise can stimulate medial-temporal neurogenesis and ameliorate cognition and symptoms/functioning in this vital group. In the proposed study, an expert team of experienced prodromal and exercise investigators will follow a group of 15 UHR adolescent and young adults (ages 16-24) through a 12 week exercise trial to determine which level of exercise intensity/frequency is tolerable for participants and optimal for improving aerobic fitness (65% of VO2max and 2 sessions per week versus 85% intensity and 3 sessions per peek) and if improvements in aerobic fitness (i.e., VO2max, VO2peak, ventilatory threshold) are associated with increases in medial temporal structure volume (hippocampus and parahippocampal gyrus) and accompanying improvements in cognitive function (i.e., including tasks known to recruit heavily on medial temporal structures) as well as symptomatology and social/role functioning. If the benchmarks are met, this data will be used to streamline a three-year rater-blind controlled trial (15 UHR-exercise, 15 UHR waitlist-control) to determine the efficacy of the intervention in promoting medial temporal health as well as accompanying cognitive, clinical, and socio-occupational function improvement. Participants will be followed up to 24-months to determine if the intervention has an affect on clinical course and transition to psychosis. Taken together, this study is important for understanding the lessons necessary for planning a future large-scale trial, and has the potential to shed light on a promising new treatment for UHR youth.

ELIGIBILITY:
Inclusion Criteria:

* age 16-24
* no history of brain injury or neurological disease
* no contraindications to exercise training (as assessed by a Clinical Translational Research Center CTRC physician)
* no history or current treatment with antipsychotics
* no contraindications for being in an magnetic resonance imaging scanner.
* meet criteria for a prodromal syndrome based upon the Structure Interview for Prodromal Syndromes (SIPS) interview.

Exclusion Criteria:

* people who are extremely claustrophobic
* have a history of significant head injury
* other physical disorder that could affect brain functioning
* mental retardation
* history of substance use disorder within 6 months of screening interview
* have a psychotic disorder (at study entry) and/or have exhibited serious self-harm behaviors
* pregnant females
* people who have contraindications to magnetic resonance (MR) scanning including intracranial, intraorbital or intraspinal metal, pacemakers, cochlear implants or other non-MR-compatible devices
* inability of the subject or their parent/guardian to understand the informed consent document
* meeting criteria for an Axis I psychotic disorder

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijay A Mittal, Ph.D., Principal Investigator — University of Colorado, Boulder; Angela Bryan, Ph.D., Principal Investigator — University of Colorado, Boulder
Locations (1):
- ADAPT Program, Boulder, Colorado, United States

REFERENCES:
- [Background] Mittal VA, Gupta T, Orr JM, Pelletier-Baldelli A, Dean DJ, Lunsford-Avery JR, Smith AK, Robustelli BL, Leopold DR, Millman ZB. Physical activity level and medial temporal health in youth at ultra high-risk for psychosis. J Abnorm Psychol. 2013 Nov;122(4):1101-10. doi: 10.1037/a0034085. PMID 24364613
- [Background] Miller TJ, McGlashan TH, Rosen JL, Cadenhead K, Cannon T, Ventura J, McFarlane W, Perkins DO, Pearlson GD, Woods SW. Prodromal assessment with the structured interview for prodromal syndromes and the scale of prodromal symptoms: predictive validity, interrater reliability, and training to reliability. Schizophr Bull. 2003;29(4):703-15. doi: 10.1093/oxfordjournals.schbul.a007040. PMID 14989408
- [Background] Niendam TA, Bearden CE, Zinberg J, Johnson JK, O'Brien M, Cannon TD. The course of neurocognition and social functioning in individuals at ultra high risk for psychosis. Schizophr Bull. 2007 May;33(3):772-81. doi: 10.1093/schbul/sbm020. Epub 2007 Apr 9. PMID 17420177
- [Background] Ragland JD, Ranganath C, Barch DM, Gold JM, Haley B, MacDonald AW 3rd, Silverstein SM, Strauss ME, Yonelinas AP, Carter CS. Relational and Item-Specific Encoding (RISE): task development and psychometric characteristics. Schizophr Bull. 2012 Jan;38(1):114-24. doi: 10.1093/schbul/sbr146. Epub 2011 Nov 28. PMID 22124089
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Patenaude B, Smith SM, Kennedy DN, Jenkinson M. A Bayesian model of shape and appearance for subcortical brain segmentation. Neuroimage. 2011 Jun 1;56(3):907-22. doi: 10.1016/j.neuroimage.2011.02.046. Epub 2011 Feb 23. PMID 21352927
- [Derived] Dean DJ, Bryan AD, Newberry R, Gupta T, Carol E, Mittal VA. A Supervised Exercise Intervention for Youth at Risk for Psychosis: An Open-Label Pilot Study. J Clin Psychiatry. 2017 Nov-Dec;78(9):e1167-e1173. doi: 10.4088/JCP.16m11365. PMID 29178684
- See also: ADAPT Program Study Site Providing Details for the Clinical Trial — http://www.adaptprogram.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 65% of V02 Max, 3x Per Week, 3 Months - Dosage/Tolerance Study: 65% of V02 Max, 3x per week, 3 months
  Exercise 1: 65% of VO2max and 2 sessions per week
  Initial study that is a separate sample from the waitlist and HIIT RCT groups
- 85% of VO2 Max, 2x Per Week, 3 Months - Study 1 Dosage: 85% of VO2 Max, 2x per week, 3 months
  Exercise 2: 85% intensity and 3 sessions per peek
  Initial tolarance study with separate participants from the RCT groups.
- Waitlist - RCT Study: Waitlist (three months no intervention) Group is a part of RCT study and a separate sample than the dosage and tolerance initial study sample.
- High Impact Interval Exercise 80%/95% VO2 Max RCT: For initial tolerance, the treadmill exercise intensity was set to elicit 55% of the participant's VO2max which was increased to 80% gradually over the first 3 weeks. During the remainder of the trial (21 weeks), the 2 weekly, treadmill sessions were designed to elicit 80% of VO2max for the majority of the time with 1-min high-intensity intervals at 95% of VO2max, every 10 minutes for 3 repetitions for a total of 30 mins. This protocol was adapted from findings in the open-label pilot study (groups 1 (65%) and 2(85%)), which suggested that fewer sessions and higher intensity of exercise were needed.
Period: Overall Study
Arm/Group | 65% of V02 Max, 3x Per Week, 3 Months - Dosage/Tolerance Study | 85% of VO2 Max, 2x Per Week, 3 Months - Study 1 Dosage | Waitlist - RCT Study | High Impact Interval Exercise 80%/95% VO2 Max RCT
Started | 7 | 5 | 20 | 18
Completed | 7 | 2 | 12 | 13
Not Completed | 0 | 3 | 8 | 5
Not completed — Withdrawal by Subject | 0 | 3 | 6 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3
Not completed — Emergence of Psychosis or Substance disorder during protocol | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Exercise - High Impact Interval 95% VO2 Max -32 Week: The exercise group participants completed a 3-month exercise treatment twice a week at moderate to intense levels of aerobic exercise (24 sessions over 12 weeks). To limit the perceived barriers to sessions,15 participants were provided with free transportation to the sessions, after the session access to healthy snacks and refreshments were provided. Participants received paid compensation after each session. All sessions were conducted as one-on-one sessions by the same exercise physiologist under the supervision of a physician to build rapport with participants and ensure consistency in the protocol. These high-intensity interval exercise sessions were tailored to the individual's exercise fitness level based on the baseline VO2max assessment. For initial tolerance, the treadmill exercise intensity was set to elicit 55% of the participant's VO2max which was increased to 80% gradually over the first 3 weeks. During the remainder of the trial (21 weeks), the 2 weekly, treadmill sessions were designed to elicit 80% of VO2max for the majority of the time with 1-min high-intensity intervals at 95% of VO2max, every 10 minutes for 3 repetitions for a total of 30 mins. This protocol was adapted from findings in the open-label pilot study, which suggested that fewer sessions and higher intensity of exercise were needed. After the exercise intervention, participants repeated the baseline visit again with separate study staff who were blinded to their exercise intervention status.
- Wait List: These individuals completed cognitive assessment, clinical assessment, and MRIs at baseline and follow up, but were not provided with exercise intervention. All assessors were blind to intervention status.
- Dosage Study 85% Vigorous: Participants were randomly assigned to 1 of 2 conditions:
  moderate or vigorous. The moderate condition required exercise 2 days a week at 65% of their Vo 2max for a total of 24 sessions. of 36 sessions. Participants wore a Polar FT1 heart rate monitor (https://www.polar.com/us-en) throughout each exercise session, and an exercise physiologist monitored the participant's exercise in order to keep the participant's heart rate at ± 5% of the prescribed target intensity. Initial exercise sessions lasted 15 minutes at 55% of Vo 2max intensity and were gradually increased to 30 minutes and target intensity within the first 3 weeks. The remaining exercise sessions lasted 30 minutes and were conducted at prescribed exercise intensity. Participants were given the choice to ride stationary bikes, run/walk on treadmills, or use elliptical machines at each session.
- Dosage Study 65%Moderate: Participants were randomly assigned to 1 of 2 conditions:
  moderate or vigorous. The moderate condition required exercise 2 days a week at 65% of their Vo 2max for a total of 24 sessions. Participants wore a Polar FT1 heart rate monitor (https://www.polar.com/us-en) throughout each exercise session, and an exercise physiologist monitored the participant's exercise in order to keep the participant's heart rate at ± 5% of the prescribed target intensity. Initial exercise sessions lasted 15 minutes at 55% of Vo 2max intensity and were gradually increased to 30 minutes and target intensity within the first 3 weeks. The remaining exercise sessions lasted 30 minutes and were conducted at prescribed exercise intensity. Participants were given the choice to ride stationary bikes, run/walk on treadmills, or use elliptical machines at each session.
- Total: Total of all reporting groups
Arm/Group | Exercise - High Impact Interval 95% VO2 Max -32 Week | Wait List | Dosage Study 85% Vigorous | Dosage Study 65%Moderate | Total
Number analyzed (Participants) | 18 | 20 | 5 | 7 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 5 | 7 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Dose study initial sample n=12; RCT study initial sample n=38, 7 withdrew (1 exercise/6 waitlist); 3 were excluded from the exercise group for not completing all 24 trials, 2 developed substance use disorders after baseline, 1 waitlist converted to a psychosis diagnosis during the protocol and was excluded, 13 withdrew/excluded in RCT; final RCT sample n=25. Across studies, 16 excluded. Final n=37.
  years
    number analyzed (Participants) | 13 | 12 | 5 | 7 | 37
    (all) | 21.15 (1.75) | 21.57 (1.78) | 19.2 (1.30) | 19.6 (1.13) | 21.36 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Dose study initial sample n=12; RCT study initial sample n=38, 7 withdrew (1 exercise/6 waitlist); 3 were excluded from the exercise group for not completing all 24 trials, 2 developed substance use disorders after baseline, 1 waitlist converted to a psychosis diagnosis during the protocol and was excluded, 13 withdrew/excluded in RCT; final RCT sample n=25. Across studies, 16 excluded. Final n=37.
  Participants
    number analyzed (Participants) | 13 | 12 | 5 | 7 | 37
    Female | 11 | 3 | 2 | 4 | 20
    Male | 2 | 9 | 3 | 3 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Dose study initial sample n=12; RCT study initial sample n=38, 7 withdrew (1 exercise/6 waitlist); 3 were excluded from the exercise group for not completing all 24 trials, 2 developed substance use disorders after baseline, 1 waitlist converted to a psychosis diagnosis during the protocol and was excluded, 13 withdrew/excluded in RCT; final RCT sample n=25. Across studies, 16 excluded. Final n=37.
  Participants
    number analyzed (Participants) | 13 | 12 | 5 | 7 | 37
    American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
    Asian | 1 | 2 | 1 | 0 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 7 | 1 | 0 | 0 | 8
    White | 3 | 8 | 3 | 7 | 21
    More than one race | 2 | 1 | 0 | 0 | 3
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — The number above reflects all enrolled (n=50); Those who completed all measures were n=37: Dose study initial sample n=12; RCT study initial sample n=38, 7 withdrew (1 exercise/6 waitlist); 3 were excluded from the exercise group for not completing all 24 trials, 2 developed substance use disorders after baseline, 1 waitlist converted to a psychosis diagnosis during the protocol and was excluded, 13 withdrew/excluded in RCT; final RCT sample n=25. Across studies, 16 excluded. Final n=37.
  participants
    United States | 18 | 20 | 5 | 7 | 50
Wide Range Achievement Test (WRAT) reading subscale [Mean (Standard Deviation); unit: Standard Score] — Population: RCT study dropout/excluded n=13; Dose study cognition was assessed with the MATRICS Consensus Cognitive Battery composite using a t-score (0=population mean, standard deviation=10), and Wide Range Achievement Test (WRAT) Reading Subscale in the RCT study using a standard score (100=population mean, standard deviation=15). On both measures, higher scores indicate better cognitive performance.
  Standard Score
    number analyzed (Participants) | 13 | 12 | 5 | 7 | 37
    (all) | 105.83 (13.38) | 114.8 (14.97) | 50.2 (7.92) | 48.5 (7.4) | 110.315 (14.17)
Relational and Item-Specific Encoding Task [Mean (Standard Deviation); unit: recollection accuracy score] — Population: RCT study dropout/excluded n=13 (see above); Dosage study working memory was assessed with the MATRICS Consensus Cognitive Battery working memory subscale using a t-score (0=population mean, standard deviation=10) and Relational and Item-Specific Encoding Task accuracy score in the RCT study using a task specific accuracy (the proportion of false alarms from the proportion of hits; range 0-100%). On both measures higher scores indicate better working memory performance.
  recollection accuracy score
    number analyzed (Participants) | 13 | 12 | 5 | 7 | 37
    (all) | 2.75 (0.45) | 3.73 (0.44) | 47.2 (6.80) | 49.7 (7.57) | 3.24 (.44)
VO2max assessment modified Balke protocol [Mean (Standard Deviation); unit: ml/kg/min] — Population: Dose study initial sample n=12; RCT study initial sample n=38, n=13 withdrew/excluded; final RCT sample n=25. Total across studies n=37. VO2 Max is calculated as ratio (mL/kg/min) during exercise; higher VO2 max indicates greater cardiovascular health.
  ml/kg/min
    number analyzed (Participants) | 13 | 12 | 5 | 7 | 37
    (all) | 33.92 (7.4) | 31.48 (8.87) | 42 (4.13) | 40.5 (4.52) | 32.7 (8.14)
Structured Interview for Psychosis-Risk Syndromes (SIPS) [Mean (Standard Deviation); unit: Symptom Severity Score] — Population: Dose study initial sample n=12; RCT study initial sample n=38, n=13 withdrew/excluded; final RCT sample n=25. Total across studies n=37. Structured Interview for Psychosis Risk Syndrome (SIPS) score is calculated as a composite of the frequency and severity of psychosis symptoms, assesses uncommon experiences there is not a relevant population reference. A higher score indicates a higher number, frequency, and/or severity of symptoms.
  Symptom Severity Score
    number analyzed (Participants) | 13 | 12 | 5 | 7 | 37
    (all) | 12.08 (3.52) | 13.50 (3.90) | 11.2 (5.89) | 13.1 (4.38) | 13.15 (3.71)

OUTCOME MEASURES:

1. Primary Outcome: Brain Volume
Description: Medial temporal structures (hippocampus and parahippocampal gyrus) will be delineated automatically using the FMRIB's Integrated Registration and Segmentation Tool algorithm within the FMRIB's Software Library (FSL) image-processing suite. Secondly, the structures will be evaluated with vertex analyses (assessing changes in shape post trial on a per-vertex basis), which will also be carried out utilizing FIRST. Shape/appearance models used in FIRST are constructed from manually segmented images provided by the Center for Morphometric Analysis (CMA, Boston). This approach is different from using a whole-structure summary measure like volume, as it allows visualization of the region of the shape that is changing as well as the type of shape change.
Time Frame: pre-trial, post-trial (3-months)
Population: Withdrew/excluded 3 Dosage (Exercise 2 group); 13 RCT (3 were excluded from the exercise group for not completing all 24 trials, 2 developed substance use disorders after baseline, 1 waitlist converted to a psychosis diagnosis during the protocol and was excluded); Final n=34; Change in hippocampal volume is reported below. On both measures negative scores indicate decreased hippocampal volumes over the study period.
Measure: Mean (Standard Deviation); unit: Change in mm cubed (baseline -followup)
Groups:
- Dosage Study Exercise: Due to small final sample size both groups are collapsed into one. 65% of V02 Max, 3x per week, 3 months
  Exercise 1: 65% of VO2max and 2 sessions per week
- Doseage Study Exercise 2: Due to small final sample size both groups are collapsed into one. 85% of VO2 Max, 2x per week, 3 months
  Exercise 2: 85% intensity and 3 sessions per peek
- RCT High Impact Interval Exercise: The exercise group participants completed a 3-month exercise treatment twice a week at moderate to intense levels of aerobic exercise (24 sessions over 12 weeks). . For initial tolerance, the treadmill exercise intensity was set to elicit 55% of the participant's VO2max which was increased to 80% gradually over the first 3 weeks. During the remainder of the trial (21 weeks), the 2 weekly, treadmill sessions were designed to elicit 80% of VO2max for the majority of the time with 1-min high-intensity intervals at 95% of VO2max, every 10 minutes for 3 repetitions for a total of 30 mins.
- RCT Wait List: Completed pre/post measures with no intervention in the intervening three months
Arm/Group | Dosage Study Exercise | Doseage Study Exercise 2 | RCT High Impact Interval Exercise | RCT Wait List
Number analyzed (Participants) | 7 | 2 | 13 | 12
Change in mm cubed (baseline -followup) | 19.8 (50.8) | 54.8 (323) | -0.489 (0.104) | -6.28 (1.95)

2. Secondary Outcome: Working Memory Assessment
Description: Working Memory Assessment - Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) battery working memory subscale - a higher score indicates working memory better performance. The Relational and Item-Specific Encoding task includes visual object representations of word stimuli. Subjects make a two-button "yes/no" response to indicate whether items in each pair had been presented "together."To prevent additional encoding of the relational object pairs the item recognition task precedes the associated recognition task. Higher scores reflect the familiarity and recollection performance as well as hit rates and false alarm rates following encoding - better performance. MATRICS Consensus Cognitive Battery working memory subscale using a t-score (0=population mean, standard deviation=10) and Relational and Item-Specific Encoding Task accuracy score in the RCT study using a task specific accuracy (d prime range; 0-100%).
Time Frame: pre-trial, post-trial (3-months)
Population: Because there were few participants who completed the vigorous condition, subsequent analyses of the exercise intervention collapsed across conditions - Exercise 1 is all exercise Pre and Exercise 2 is all exercise post - Arm 2 has pre/Post for intervention group and wait list group listed for the RISE measure
Measure: Mean (Standard Deviation); unit: Composite tscore/ RiSE Score
Groups:
- Pre-Intervention 85% Dosage Study: 85% of V02 Max, 3x per week, 3 months
  Exercise 1: 65% of VO2max and 2 sessions per week
- Post-Intervention Dosage Study: 85% of VO2 Max, 2x per week, 3 months Exercise 2: 85% intensity and 3 sessions per peek
- RCT Exercise Pre-Intervention; RCT Exercise Post-Intervention: In this group the treadmill exercise intensity was set to elicit 55% of the participant's VO2max which was increased to 80% gradually over the first 3 weeks. During the remainder of the trial (21 weeks), the 2 weekly, treadmill sessions were designed to elicit 80% of VO2max for the majority of the time with 1-min high-intensity intervals at 95% of VO2max, every 10 minutes for 3 repetitions for a total of 30 mins
- RCT Waitlist Pre-Intervention: This is the baseline measure of the group with no exercise intervention.
- RCT Waitlist Post-Intervention Period: This is the group with no exercise intervention 3 months later.
- Pre-Intervention Moderate Dosage - 65%: 65% of V02 Max, 3x per week, 3 months
  Exercise 1: 65% of VO2max and 2 sessions per week
- Post-Intervention Moderate Dosage - 65%: 65% of V02 max , 3 x per week 3 months
Arm/Group | Pre-Intervention 85% Dosage Study | Post-Intervention Dosage Study | RCT Exercise Pre-Intervention | RCT Exercise Post-Intervention | RCT Waitlist Pre-Intervention | RCT Waitlist Post-Intervention Period | Pre-Intervention Moderate Dosage - 65% | Post-Intervention Moderate Dosage - 65%
Number analyzed (Participants) | 2 | 2 | 13 | 13 | 13 | 13 | 7 | 7
Composite tscore/ RiSE Score | 47.5 (14.8) | 53 (19.8) | 2.75 (.45) | 3.00 (.57) | 3.73 (.44) | 3.13 (.56) | 48.5 (7.40) | 52.9 (6.91)

3. Other Pre Specified Outcome: Attenuated Psychosis Positive Symptom Subscales
Description: The Structured Interview for Prodromal Symptoms (SIPS) will be administered to formally assess attenuated positive symptoms after inclusion in the study. It will also be administered post-trial to track changes in clinical symptoms post intervention trial. The SIPS rates the severity of relevant dimensions including positive symptoms along a 7-point scale ranging from absent (0) to severe and psychotic (6) across five symptom categories, resulting in a score that ranges from 0 (no positive symptoms) to 30 (psychosis along all symptoms dimensions).
Time Frame: pre-trial, post-trial (3-months)
Population: Withdrew/excluded 3 Dosage (85% VO2 Max group); 13 RCT (3 were excluded from the exercise group for not completing all 24 trials, 2 developed substance use disorders after baseline, 1 waitlist converted to a psychosis diagnosis during the protocol and was excluded); Final n=34
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre Intervention - Moderate Dosage - 65% V02 Max: 65% of V02 Max, 3x per week, 3 months
  Exercise 1: 65% of VO2max and 2 sessions per week
- Post Intervention - Moderate Dosage - 65% V02 Max: 65% of VO2 Max, 2x per week, 3 months 65% intensity and 3 sessions per peek
- RCT Waitlist: In this group the treadmill exercise intensity was set to elicit 55% of the participant's VO2max which was increased to 80% gradually over the first 3 weeks. During the remainder of the trial (21 weeks), the 2 weekly, treadmill sessions were designed to elicit 80% of VO2max for the majority of the time with 1-min high-intensity intervals at 95% of VO2max, every 10 minutes for 3 repetitions for a total of 30 mins.
- RCT Exercise Post-Intervention: This group experienced no exercise intervention over the 3 month period.
- RCT Waitlist Post-Intervention: This group experienced no exercise intervention during the 3 month study period.
- Pre-Intervention Vigorous Dosage Condition Vigorous Dosage- 85% of V02 Max; Post-Intervention - Vigorous Dosage Condition -85 % VO2 Max: 85% of VO2 Max, 2x per week, 3 months
  Exercise 2: 85% intensity and 3 sessions per peek
Arm/Group | Pre Intervention - Moderate Dosage - 65% V02 Max | Post Intervention - Moderate Dosage - 65% V02 Max | RCT Exercise Pre-Intervention | RCT Waitlist | RCT Exercise Post-Intervention | RCT Waitlist Post-Intervention | Pre-Intervention Vigorous Dosage Condition Vigorous Dosage- 85% of V02 Max | Post-Intervention - Vigorous Dosage Condition -85 % VO2 Max
Number analyzed (Participants) | 7 | 7 | 13 | 12 | 13 | 12 | 2 | 2
score on a scale | 13.1 (4.38) | 9.29 (3.82) | 12.08 (3.52) | 13.50 (3.90) | 8 (3.46) | 11.38 (3.82) | 14 (8.49) | 12 (5.66)

4. Other Pre Specified Outcome: Aerobic Fitness
Description: VO2max was assessed via a modified Balke protocol by an exercise physiologist under the supervision of a physician. In this modified Balke protocol, the treadmill speed was individualized in a procedure to elicit 70% of the age-predicted max heart rate and ratings of a "somewhat hard" perceived exertion (RPE). Then, the speed of the treadmill remained the same throughout the test, but the incline of the treadmill belt increased 2% every 2 min (or 2.5% for speeds 6 mph or greater) to exhaustion. Tests generally lasted 8-12 minutes to attain the recommended target for VO2max testing. Measures indicate cardiovascular health with higher scores indicating greater health.
Time Frame: pre-trial, post-trial (3 months)
Population: Because there were few participants (n=9); outcome data combine moderate (n=2) & vigorous (n=7) groups; total outcome sample n=9; 13 RCT (3 were excluded from the exercise group for not completing all 24 trials, 2 developed substance use disorders after baseline, 1 waitlist converted to a psychosis diagnosis during the protocol and was excluded); Final n=34
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Pre-Intervention- Moderate Dosage -65% VO2max: 65% of V02 Max, 3x per week, 3 months Exercise 1: 65% of VO2max and 2 sessions per week
  85% of VO2 Max, 2x per week, 3 months Exercise 2: 85% intensity and 3 sessions per peek
- Post-Intervention- Moderate Dosage -65% VO2max: 65% of V02 Max, 3x per week, 3 months Exercise 1: 65% of VO2max and 2 sessions per week
- Pre-Intervention - Vigorous Dosage; Post-Intervention Vigorous Exercise - 85% VO2max: 85% of VO2 Max, 2x per week, 3 months Exercise 2: 85% intensity and 3 sessions per peek
- RCT: Exercise Pre-Intervention; RCT: Exercise Post-Intervention: This exercise group completed a 3-month exercise treatment twice a week at moderate to intense levels of aerobic exercise (24 sessions over 12 weeks). To limit the perceived barriers to sessions,15 participants were provided with free transportation to the sessions, after the session access to healthy snacks and refreshments were provided. Participants received paid compensation after each session. All sessions were conducted as one-on-one sessions by the same exercise physiologist under the supervision of a physician to build rapport with participants and ensure consistency in the protocol. These high-intensity interval exercise sessions were tailored to the individual's exercise fitness level based on the baseline VO2max assessment. For initial tolerance, the treadmill exercise intensity was set to elicit 55% of the participant's VO2max which was increased to 80% gradually over the first 3 weeks. During the remainder of the trial (21 weeks), the 2 weekly, treadmill sessions were designed to elicit 80% of VO2max for the majority of the time with 1-min high-intensity intervals at 95% of VO2max, every 10 minutes for 3 repetitions for a total of 30 mins.
- RCT: Wait List Pre-Intervention Period; RCT: Wait List Post-Intervention Period: Completed Baseline and follow up measures with no intervening intervention
Arm/Group | Pre-Intervention- Moderate Dosage -65% VO2max | Post-Intervention- Moderate Dosage -65% VO2max | Pre-Intervention - Vigorous Dosage | Post-Intervention Vigorous Exercise - 85% VO2max | RCT: Exercise Pre-Intervention | RCT: Exercise Post-Intervention | RCT: Wait List Pre-Intervention Period | RCT: Wait List Post-Intervention Period
Number analyzed (Participants) | 7 | 7 | 2 | 2 | 13 | 13 | 12 | 12
ml/kg/min | 40.5 (10.9) | 39.0 (10.1) | 40.2 (6.15) | 41.2 (0.495) | 33.92 (7.4) | 38.2 (7.8) | 31.48 (7.8) | 32.97 (7.2)

ADVERSE EVENTS:
Time Frame: No exercise intervention related or adjacent events were recorded during the trials period (12 weeks), despite clinical and exercise physiologist assessment. Dose study (moderate intensity) assessed 2x a week for 12 weeks; dose study (high intensity) assessed 3x a week for 12 weeks; RCT assessed 2x a week for 12 weeks; waitlist group assessed at baseline and 3-month follow-up.
Description: No exercise exercise intervention related or adjacent events were recorded during the trials period (12 weeks), despite clinical and exercise physiologist assessment.
  Withdrew/excluded 3 Dosage (85% VO2 Max group); 13 RCT (3 were excluded from the exercise group for not completing all 24 trials, 2 developed substance use disorders after baseline, 1 waitlist converted to a psychosis diagnosis during the protocol and was excluded); Final n=34
Groups:
- Dosage Study: Exercise - Moderate Intensity: The moderate condition required exercise 2 days a week at 65% of their Vo2max for a total of 24 sessions.
  Adverse potential events were exercise related injury which were assessed by an exercise physiologist during bi-weekly interventions.
- Dosage Study: Exercise High Intensity: The vigorous condition required exercise 3 days a week at 85% of the participant's Vo2max for a total of 36 sessions.
  Adverse potential events were exercise related injury which were assessed by an exercise physiologist during bi-weekly interventions.
- RCT: Exercise - High Impact Interval 95%/80% VO2 Max -32 Week: The exercise group participants completed a 3-month exercise treatment twice a week at moderate to intense levels of aerobic exercise (24 sessions over 12 weeks). For initial tolerance, the treadmill exercise intensity was set to elicit 55% of the participant's VO2max which was increased to 80% gradually over the first 3 weeks. During the remainder of the trial (21 weeks), the 2 weekly, treadmill sessions were designed to elicit 80% of VO2max for the majority of the time with 1-min high-intensity intervals at 95% of VO2max, every 10 minutes for 3 repetitions for a total of 30 mins.32 This protocol was adapted from findings in the open-label pilot study, which suggested that fewer sessions and higher intensity of exercise were needed. 7 After the exercise intervention, participants repeated the baseline visit again with separate study staff who were blinded to their exercise intervention status.
  Adverse potential events were exercise related injury which were assessed by an exercise physiologist during bi-weekly interventions.
- RCT: Wait List: These individuals completed cognitive assessment, clinical assessment, and MRIs at baseline and follow up, but were not provided with exercise intervention. All assessors were blind to intervention status.
  No adverse potential events related to exercise related injury were anticipated in the waitlist group. Assessment occurred at baseline and 3-month follow-up.
Arm/Group | Dosage Study: Exercise - Moderate Intensity | Dosage Study: Exercise High Intensity | RCT: Exercise - High Impact Interval 95%/80% VO2 Max -32 Week | RCT: Wait List
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/7 | 0/2 | 0/13 | 0/12

LIMITATIONS AND CAVEATS:
It is a notable limitation that the current sample size is small; however, the current sample size is comparable or larger than extant randomized control studies in psychosis CHR-p individuals make up a heterogenous population future studies should consider heterogeneity in clinical and cognitive symptoms in larger samples. There are several benefits of exercise not examined by the current study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT02155699/Prot_SAP_000.pdf